CLINICAL TRIAL: NCT02585596
Title: A Double-blind, Randomized, Parallel, Placebo-active Controlled, Multi-center Phase II Clinical Trial to Investigate the Efficacy and Safety of YH23537 Following 12-week Oral Administration in Patients With Chronic Periodontal Disease
Brief Title: A Phase II Clinical Trial of YH23537 in Patients With Chronic Periodontal Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YH23537-201
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- YH23537 1000mg/day (Experimental): YH23537 500mg 1 tab, placebo 500mg 2tab twice a day (before morning,evening meal) during 12 weeks
  Interventions: Drug: YH23537 1000mg/day; Drug: placebo
- YH23537 2000mg/day (Experimental): YH23537 500mg 2tab, placebo 500mg 1tab twice day (before morning,evening meal) during 12 weeks
  Interventions: Drug: YH23537 2000mg/day; Drug: placebo
- YH23537 3000mg/day (Experimental): YH23537 500mg 3tab a day twice day (before morning,evening meal) during 12 weeks
  Interventions: Drug: YH23537 3000mg/day
- YH23537 3000mg/day loading 1000mg/day (Experimental): YH23537 500mg 3tab twice a day (before morning,evening meal) during 4weeks and YH23537 500mg tab twice a day (before morning,evening meal) during 8weeks
  Interventions: Drug: YH23537 1000mg/day; Drug: YH23537 3000mg/day; Drug: placebo
- Placebo (Placebo Comparator): YH23537 500mg placebo 3tab twice a day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: YH23537 1000mg/day — YH23537 500mg 2 tab
  Arms: YH23537 1000mg/day; YH23537 3000mg/day loading 1000mg/day
Drug: YH23537 2000mg/day — YH23537 500mg 4 tab
  Arms: YH23537 2000mg/day
Drug: YH23537 3000mg/day — YH23537 500mg 6 tab
  Arms: YH23537 3000mg/day; YH23537 3000mg/day loading 1000mg/day
Drug: placebo — YH23537 500mg tab placebo
  Arms: Placebo; YH23537 1000mg/day; YH23537 2000mg/day; YH23537 3000mg/day loading 1000mg/day

SUMMARY:
This study is designed to evaluate the efficacy and the safety of YH23537 in Korea patients with chronic periodontitis, in order to investigate the recommended therapeutic dose.

DETAILED DESCRIPTION:
at screening visit, at least existing 18 teeth,Mild/moderate/severe periodontitis patients diagnosed with chronic periodontitis according to the CDC / AAP (Center for Disease Control / American Academy for Periodontology) periodontitis classification (2012).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 19 years of age or older
* Have at least 18 natural teeth
* have been diagnosed with chronic periodontitis
* have been diagnosed Mild/Moderate/Severe periodontitis with according to CDC / AAP periodontal classification (2012))
* Provide informed consent and willingness to cooperate with the study protocol

Exclusion Criteria:

* Women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study and for up to 4 weeks after the last dose of investigational product.
* Pregnant or lactating females
* Systemic diseases such as diabetes and hypertension
* Patients who take Anticoagulants or Antiplatelet Agents
* Continually use for phenytoin, calcium channel blocker, cyclosporin, coumarin, nonsteroidal anti-inflammatory drugs and aspirin use in the previous one month
* Patients who received periodontal treatment within the last 6 months
* Patients who have malignant tumor
* History of positive serologic evidence of current infectious liver disease including HbsAg, or anti-HCV.
* Patients with mental retardation and dementia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Change in probing pocket depth (PD) | baseline, 4weeks, 8week, 12weeks

SECONDARY OUTCOMES:
Change in Clinical attachment level (CAL) | baseline, 4weeks, 8week, 12weeks
Change in Bleeding on probing(BOP) | baseline, 4weeks, 8week, 12weeks
Change in Gingival recession(GR) | baseline, 4weeks, 8week, 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Incheol Rhyu, Ph.D., Study Chair — Seoul National University Hospital
Locations (1):
- Incheol Rhyu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No